CLINICAL TRIAL: NCT01391026
Title: Computer Assisted Quality of Life and Symptom Assessment of Complex Patients
Brief Title: Computer Assisted Symptom Evaluation of Complex Patients
Acronym: CASE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cook County Health (Other Government)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Principal Investigator, William Trick, Principal Investigator, Cook County Health
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 10-143; 1R24HS019481-01 (AHRQ)
Record Dates: First submitted 2011-07-07; First posted 2011-07-11 (Estimated); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Multiple Co-morbidities
Keywords: Medical informatics; Health services accessibility

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Usual care (No Intervention): Patients will receive usual care by their primary care physicians without automated referral to specialized providers.
- Enhanced patient-centered care (Experimental): Patients will be evaluated and treated in the advanced illness management clinic
  Interventions: Behavioral: Enhanced patient-centered care

INTERVENTIONS:
Behavioral: Enhanced patient-centered care — The experimental arm will be referred to a multi-disciplinary clinic
  Arms: Enhanced patient-centered care

SUMMARY:
Patients who have advanced or multiple chronic illnesses present management difficulties for primary care providers. Acute medical issues and limited time for patient evaluation can complicate complete assessment of physical symptoms that directly impact a patient's quality of life. The Cook County Health and Hospitals System (CCHHS) established an Advanced Illness Management Clinic to provide care for complex patients. Patient entry into the Advanced Illness Management Clinic is by referral only, a passive process. After discharge, general medicine clinic patients who do not have a medical provider are given an appointment in the clinic. Since the hospital is the source of many patients, this guarantees that these patients will have at least one illness advanced enough to require hospitalization, and most will have additional chronic illnesses. An outpatient palliative care clinic located in a specialty clinic setting was initiated in 2004. The goal of the clinic was to extend the benefits realized by hospital patients, for whom palliative care consultation has been available for many years, to patients cared for in the outpatient setting. The benefits provided include physical symptom management, spiritual counseling, and support for social issues. Until recently, this outpatient palliative care model has mainly served patients with malignancy. With the addition of the Advanced Illness Management Clinic, palliative care clinicians now can provide care to patients with other chronic and serious illness in the primary care setting.

Hypothesis: Complex patients will have improved quality of life and a reduced symptom burden if seen by a multidisciplinary clinic post-hospitalization, compared to usual care in a general medicine clinic.

DETAILED DESCRIPTION:
Outcome measures:

1. Quality of life as measured by the National Institutes of Health (NIH) Patient Reported Outcomes Measurement Information System (PROMIS) short form
2. Physical symptom burden as measured by the Memorial Symptom Assessment Scale (MSAS), short form

ELIGIBILITY:
Inclusion Criteria:

* English or Spanish speaker
* Must be a general medicine clinic patient
* Must have a physical symptom score on MSAS above threshold (i.e., 1.0 or higher)
* Must have a phone number for contact

Exclusion Criteria:

* Visual or cognitive impairment

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2011-06; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
NIH PROMIS 10-item short form quality of life | 6 months
  We will assess the physical and mental components of the quality of life instrument

SECONDARY OUTCOMES:
MSAS physical symptom score | 6 months
Healthcare utilization | 6 months
  We will monitor healthcare utilization within our system. To include visits to the emergency room, clinics, and hospitalizations.

CONTACTS AND LOCATIONS:
Overall Officials: William E Trick, MD, Principal Investigator — Cook County Health & Hospitals System
Locations (1):
- Stroger Hospital of Cook County, Chicago, Illinois, United States